CLINICAL TRIAL: NCT04996953
Title: The Correlation Study of Hypnotic Drugs on the Cognitive Function of Patients With Chronic Insomnia.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Lili Cao (Other)
Responsible Party: Sponsor-Investigator, Lili Cao, Professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: KUN0802
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Insomnia Chronic
Keywords: Insomnia; Cognitive disorder; Hypnotic; Memory
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 165 patients with insomnia

SUMMARY:
All the subjects were assessed for sleep quality, anxiety and depression, and cognitive function. Based on their previous hypnotic medication history, they were divided into a non-medicine group and a benzodiazepine group，and the group taking non-benzodiazepine drugs.The cognitive effects of different hypnotic drugs on patients were evaluated by comparing sleep related scale and cognitive function scale.

DETAILED DESCRIPTION:
Insomnia is one of the most common sleep disorders, with 38.2% of Chinese people suffering from sleep disorders. There are many ways to treat insomnia disorders, but drug therapy is the most commonly used method by medical staff. The cognitive effects of sleep drugs vary in numerous studies, depending on the type and dosage of drugs.This study aims to explore the effects of different types of hypnotic drugs on the treatment of insomnia and cognitive function, hoping to improve the sleep quality and living standards of insomnia patients through this study, and also to obtain some cognitive impairment prevention measures related to insomnia, to provide some theoretical basis for clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent, male or female ≥18 and ≤75 years old;
2. (ICSD-3) proposed the diagnostic criteria for chronic insomnia;

2. Did not take hypnotic drugs before the visit; 3. Those who took hypnotic drugs before the visit; 4. Can understand and comply with the study protocol;

Exclusion Criteria:

1. Severe organic disease;
2. Any suicidal behavior in the past 10 years;
3. Those who cannot communicate normally cannot cooperate to complete the scale test;
4. Women who are breastfeeding or pregnant;
5. Medical history that the investigator believes could affect the safety of the subject or interfere with the study evaluation;
6. Currently diagnosed with sleep apnea, narcolepsy and other sleep disorders;
7. Sleep disorders caused by central nervous system diseases, or neurodegenerative diseases such as Parkinson's disease, Alzheimer's disease, lewy bodies dementia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects were patients in the outpatient department of Qianfoshan Hospital in Shandong Province from August 2019 to June 2025. All patients met the diagnostic criteria for chronic insomnia.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index scale | 1 day
  The sleep quality of the patients in the past month was evaluated. The higher the score, the worse the sleep quality. The scale of the score is 0-21, and the higher score means a worse outcome.
Epworth Sleeping Scale | 1 day
  Assess the possibility of dozing (not just feeling tired) in recent months. The higher the score was, the more likely it was to doze during the day. The scale of the score is 0-24, and the higher score means a worse outcome.
Insomnia Severity Index | 1 day
  Liker scale is used to evaluate the nature and symptoms of sleep disorders. The higher the score, the more serious the insomnia. The scale of the score is 0-28, and the higher score means a worse outcome.
Hamilton Anxiety Scale | 1 day
  It can be used to evaluate the depressive symptoms of depression, manic depression, neurosis and other diseases. The scale of the score is 0-56, and the higher score means a worse outcome.
Hamilton Depression Scale | 1 day
  It can be used to evaluate the depressive symptoms of depression, manic depression, neurosis and other diseases. The higher the score, the more severe the depression. The scale of the score is 0-96, and the higher score means a worse outcome.
The Word Learning Scale | 1 day
  used to evaluate the subjects from two aspects of immediate recall and long-term delayed recall. The evaluation content included 15 words in five categories: body parts, animals, tools, vehicles and furniture. The 15 words were first presented three times.The score of immediate recall was the total number of words recalled three times, and the score of short-term delay recall was the correct number of free recall after 2min.Among them, immediate memory lower than 18 indicates that immediate memory function is impaired, and delayed memory lower than 6 indicates that delayed memory is impaired.the higher scores mean a better outcome.
The verbal Fluency Scale | 1 day
  They were asked to name as many animals, fruits and vegetables as possible in a 60-second experiment,the higher scores mean a better outcome.
The Numeral-Sign Conversion Test Scale | 1 day
  The tester placed the test in front of the subject, with a number above it and a symbol below it, with a different symbol for each number.Subjects were given 90 seconds to fill each space with a symbol that matched the sample, and were given one point for each symbol that matched, the higher the score, the better.
Digital Span Test Scale | 1 day
  To assess the subjects' attention span, forward and backward number spans were the subjects' ability to recite a series of numbers in the correct order.Participants were asked to repeat a series of random numbers in reverse order, reading each number for one second.Participants were asked to repeat the number in reverse order.Each set of numbers was randomly composed of the numbers 1 to 9, and the highest success score was calculated.The most successful scores were back-to-back 10 points and back-to-back 8 points.The higher the score, the better.
Stroop Color Word Test Scale | 1 day
  The executive ability of the subjects was assessed by the number of questions correctly answered by the subjects within 1min, which was divided into three types of cards: A, B and C, and each card had 100 items.Subjects correctly read the total number of red, blue, and green color names printed in black on card A within 1min, correctly identify the total number of red, blue, and green color backgrounds on card B within 1min, and correctly read the total number of different colors with red, blue, and green names on card C within 1min.For all parts of the Stroop test, the result is the time required to complete the C-card task, and the correct number, which is a kind of executive function test.The longer it takes, the worse the result, the higher the correct number, the better.
Trail Making Test A and B Scale | 1 day
  Test A: Show the numbers from 1 to 25. They are randomly distributed. Connect them in the order of 1, 2, 3, all the way to 25.Test B: There are numbers 1 to 13, black and white, respectively, in the order of the color black and white cameras, such as white 1 with black 1, black 1 with white 2, white 2 with black 2, all the way to 13.the higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No